CLINICAL TRIAL: NCT05899972
Title: Study of the Influence of an Osteopathic Treatment Protocol on the Improvement of Sleep: a Double-blind Randomized Controlled Trial
Brief Title: Influence of an Osteopathic Treatment Protocol on the Improvement of Sleep Quality in Young Adults With Insomnia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Escola Superior de Tecnologia da Saúde do Porto (Other)
Responsible Party: Principal Investigator, Natália Maria Oliveira Campelo, Professor, Escola Superior de Tecnologia da Saúde do Porto
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: OST1-007
Record Dates: First submitted 2023-05-31; First posted 2023-06-12 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-04

CONDITIONS: Healthy
Keywords: Osteopathy; Insomnia; Sleep disorder
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Sleep Wake Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: In the distribution of the volunteers to the groups, the participants chose between two numbered envelopes, opaque and sealed, in order to guarantee the confidentiality of the allocation, to which group they belonged. Inside each envelope is a piece of paper with the group, control group or intervention group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Experimental group (Experimental): The protocol is initiated by the suboccipital inhibition technique, with an average duration of three minutes. Afterwards, the frontal lift and parietal lift techniques were performed, which lasted an average of five minutes, being two and a half minutes for each one. Finally, the IV ventricle technique was performed, with an average duration of three minutes.
  Interventions: Other: Suboccipital inhibition technique; Other: Frontal lift technique; Other: Parietal lift technique; Other: IV ventricle technique
- Control group (Placebo Comparator): For the control group the placebo technique will be applied for 6 minutes.
  Interventions: Other: Placebo technique

INTERVENTIONS:
Other: Placebo technique — With the volunteer in a supine position, the researcher placed the palms of their hands on the patient's shoulders. The contact is made with the hands on the shoulder blades of the volunteer for 6 minutes.
  Arms: Control group
Other: Suboccipital inhibition technique — With the volunteer in a supine position, the investigator is sitting position at the patient's bedside. The investigator starts by placing both hands under the patient's head in the occipital region. After palpating the suboccipital muscles, the investigator uses the second, third and fourth fingers of both hands flexed against the muscle belly and remains in this position.
  Arms: Experimental: Experimental group
Other: Frontal lift technique — With the volunteer in a supine position, the investigator is sitting position at the patient's bedside. The investigator positions the tips of both index fingers on either side of the metopic suture while the third finger remains resting on the frontal bone so that the tips of the fourth fingers contact the zygomatic processes bilaterally. A slight pressure is applied with the index fingers and an anterior pressure is performed.
  Arms: Experimental: Experimental group
Other: Parietal lift technique — With the volunteer in a supine position, the investigator is sitting position at the patient's bedside. The investigator places the palms on the lateral edges of the parietal bones and the thumbs crossed at the sagittal suture. First, a medial pressure is administered with the second, third and fourth fingers and then a cephalic traction is performed.
  Arms: Experimental: Experimental group
Other: IV ventricle technique — With the volunteer in a supine position, the investigator is sitting position at the patient's bedside. The investigator positions his hands in a shell and thumbs together at the level of the spinous apophyses of the patient's second or third cervical vertebra.
  Arms: Experimental: Experimental group

SUMMARY:
Sleep deprivation, which is a universal necessity, has serious physiological consequences.

Sleep disorders are among the most common health problems, and yet they are often neglected. The osteopathic treatment results in vasodilation, muscle relaxation and increased blood flow, resulting in improved range of motion, decreased pain perception and/or tissue changes. Thus, osteopathy ensures improved physical and mental health, which consequently helps patients with their sleep disorders.

DETAILED DESCRIPTION:
Humans spend about a third of their lives sleeping, but most individuals know little about sleep. Sleep deprivation, which is a universal necessity, has serious physiological consequences.

Based on behavioral and physiological criteria, human sleep is divided into two phases: Non Rapid Eye Movement (NREM) and Rapid Eye Movement (REM).

NREM sleep corresponds to 75% to 80% of sleep and REM approximately 20% to 25% of sleep, existing between four to six episodes.

Sleep disorders are among the most common health problems, and yet they are often neglected. It is estimated that millions of people suffer chronically from a sleep or wakefulness disorder, impairing their health and longevity.

According to the International Classification of Sleep Disorders (ICSD) there are eight categories of sleep disorders and clinical history is essential for diagnosis, including family history, medical, psychiatric, neurological or substance abuse disorders.

Insomnia is a sleep disorder defined by difficulty falling asleep, staying asleep, or both. It can cause significant distress and impair daily tasks. The symptoms of insomnia are expressed by having difficulty falling asleep, waking up frequently during the night, waking up very early on a daily basis, and tiredness already present upon waking up.

Osteopathic treatment results in vasodilation, muscle relaxation and increased blood flow, resulting in improved range of motion, decreased pain perception and/or tissue changes (Henley, Ivins, Mills, Wen, & Benjamin, 2008). Thus, osteopathy ensures improved physical and mental health, which consequently helps patients with their sleep disorders.

ELIGIBILITY:
Inclusion Criteria:

* Have sleep disorders (insomnia);
* Volunteers between 18 and 30 years of age.

Exclusion Criteria:

* Attending the 3rd or 4th year of the Osteopathy Course;
* Present fever (axillary or oral temperature higher than 37.5º C);
* Have a history of skull fracture;
* Have a history of bleeding and intracranial hemorrhage;
* Have a diagnosis of convulsion.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Sleep Quality assessed with the Pittsburgh Sleep Quality Index | 7 days post-intervention
  The Pittsburgh Sleep Quality Index (PSQI) is a self-report questionnaire that assesses sleep quality, measures several different aspects of sleep.

CONTACTS AND LOCATIONS:
Overall Officials: Natália MO Campelo, PhD, Principal Investigator — Escola Superior de Saúde do Politécnico do Porto
Locations (1):
- Escola Superior da Saúde do Porto, Porto, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] K Pavlova M, Latreille V. Sleep Disorders. Am J Med. 2019 Mar;132(3):292-299. doi: 10.1016/j.amjmed.2018.09.021. Epub 2018 Oct 4. PMID 30292731
- [Background] McArdle N, Ward SV, Bucks RS, Maddison K, Smith A, Huang RC, Pennell CE, Hillman DR, Eastwood PR. The prevalence of common sleep disorders in young adults: a descriptive population-based study. Sleep. 2020 Oct 13;43(10):zsaa072. doi: 10.1093/sleep/zsaa072. PMID 32280974
- [Background] Perdereau-Noel M, Saliou P, Vic P. [Prevalence of teenage sleeping disorders]. Arch Pediatr. 2017 Apr;24(4):336-345. doi: 10.1016/j.arcped.2017.01.009. Epub 2017 Feb 24. French. PMID 28242150
- [Background] Bruce ES, Lunt L, McDonagh JE. Sleep in adolescents and young adults. Clin Med (Lond). 2017 Oct;17(5):424-428. doi: 10.7861/clinmedicine.17-5-424. PMID 28974591
- [Background] Hirshkowitz M. Normal human sleep: an overview. Med Clin North Am. 2004 May;88(3):551-65, vii. doi: 10.1016/j.mcna.2004.01.001. No abstract available. PMID 15087204
- [Background] van de Wouw E, Evenhuis HM, Echteld MA. Prevalence, associated factors and treatment of sleep problems in adults with intellectual disability: a systematic review. Res Dev Disabil. 2012 Jul-Aug;33(4):1310-32. doi: 10.1016/j.ridd.2012.03.003. Epub 2012 Mar 30. PMID 22502859
- [Background] Del Rio Joao KA, Becker NB, de Neves Jesus S, Isabel Santos Martins R. Validation of the Portuguese version of the Pittsburgh Sleep Quality Index (PSQI-PT). Psychiatry Res. 2017 Jan;247:225-229. doi: 10.1016/j.psychres.2016.11.042. Epub 2016 Nov 28. PMID 27923147
- [Background] Medalie L, Cifu AS. Management of Chronic Insomnia Disorder in Adults. JAMA. 2017 Feb 21;317(7):762-763. doi: 10.1001/jama.2016.19004. No abstract available. PMID 28241342
- [Background] Chigome, Audrey & Nhira, Sandra & Meyer, Johanna. (2018). An overview of insomnia and its management. SA Pharmaceutical Journal. 85. 32-38.
- [Background] Cutler MJ, Holland BS, Stupski BA, Gamber RG, Smith ML. Cranial manipulation can alter sleep latency and sympathetic nerve activity in humans: a pilot study. J Altern Complement Med. 2005 Feb;11(1):103-8. doi: 10.1089/acm.2005.11.103. PMID 15750368
- [Background] Henley CE, Ivins D, Mills M, Wen FK, Benjamin BA. Osteopathic manipulative treatment and its relationship to autonomic nervous system activity as demonstrated by heart rate variability: a repeated measures study. Osteopath Med Prim Care. 2008 Jun 5;2:7. doi: 10.1186/1750-4732-2-7. PMID 18534024
- [Background] Byun JI, Shin YY, Chung SE, Shin WC. Safety and Efficacy of Gamma-Aminobutyric Acid from Fermented Rice Germ in Patients with Insomnia Symptoms: A Randomized, Double-Blind Trial. J Clin Neurol. 2018 Jul;14(3):291-295. doi: 10.3988/jcn.2018.14.3.291. Epub 2018 Apr 27. PMID 29856155
- [Background] Nobles, T., Bach, A., & Boesler, D. (2016). Case report of osteopathic treatment of insomnia and traumatic anhidrosis. International Journal of Osteopathic Medicine, 21, 58-61. https://doi.org/10.1016/j.ijosm.2016.01.006
- [Background] Hasan F, Tu YK, Yang CM, James Gordon C, Wu D, Lee HC, Yuliana LT, Herawati L, Chen TJ, Chiu HY. Comparative efficacy of digital cognitive behavioral therapy for insomnia: A systematic review and network meta-analysis. Sleep Med Rev. 2022 Feb;61:101567. doi: 10.1016/j.smrv.2021.101567. Epub 2021 Nov 10. PMID 34902820